CLINICAL TRIAL: NCT05804877
Title: Efficacy of an Online Mindfulness-based Cognitive Skills Program on Depressive Symptoms and Quality of Life in University Students
Brief Title: Online MBCT Program for University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Yun-Ling Chen, Assistant Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS1-22150
Record Dates: First submitted 2023-03-05; First posted 2023-04-07 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Depression in Adolescence
Keywords: university student; online program; MBCT; depression; quality of life
MeSH Terms: conditions — Depression | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- online mindfulness-based cognitive therapy program (Experimental): The online mindfulness-based cognitive program was delivered on the platform of LINE to the experimental group 3 times a week for 8 weeks
  Interventions: Behavioral: mindfulness-based cognitive therapy
- mental health education (Placebo Comparator): The mental health education was delivered on the platform of LINE to the control group 3 times a week for 8 weeks
  Interventions: Other: Mental health education

INTERVENTIONS:
Behavioral: mindfulness-based cognitive therapy — Participants in the experimental group would be arranged to attend online mindfulness-based cognitive programs for eight weeks. Each week was divided into 3 parts, which were detailed mindfulness-based skills training with pictures or short videos, techniques application in different scenarios, and concepts consolidation through a web-based assignment.
  Arms: online mindfulness-based cognitive therapy program
Other: Mental health education — The mental health education was delivered on the platform of LINE to the control group 3 times a week for 8 weeks
  Arms: mental health education

SUMMARY:
The goal of this interventional study is to examine the efficacy of the online mindfulness-based cognitive therapy program(MBCT) in youth (18-25 years old) with depressive symptoms. The main questions it aims to answer are:

* Whether the program could reduce depressive symptoms in university students.
* Whether the program could increase quality of life in university students.
* The effectiveness, acceptance, and practicability of the program for university students.

Participants in the experimental group would be arranged to attend online mindfulness-based cognitive programs for eight weeks. The control group would be educated the knowledge of mental health to manage their negative emotions.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) was conducted to examine the efficacy of the online mindfulness-based cognitive therapy program(MBCT) in youth (18-25 years old) with depressive symptoms. The investigators expect the online MBCT program could assist university students in reducing their depressive mood and facilitating quality of life. The investigators also discussed the effectiveness, acceptance, and practicability of the online MBCT program to the subjects.

Participants in the experimental group would be arranged to attend online mindfulness-based cognitive programs for eight weeks. Each week was divided into 3 parts: detailed skill training with pictures or short videos, techniques application in different scenarios, and concepts consolidation through a web-based assignment. Participants were requested to complete the 3 parts above, which would take approximately 15 minutes in total per week. The content of the online intervention includes 8 chapters reflecting multiple topics (e.g. explaining MBCT, automatic pilot, awareness of mood, accentedness, staying with the present experience, linking habitual reactions to the unpleasant event, using breathing and body as an anchor, and planning to continue mindfulness practice) which were delivered to subjects each week by the research team.

Participants in the control group would acquire knowledge of mental health to manage their negative emotions. There would be 2 times of mental health education and one web-based assignment including writing feedback to ensure learning effectiveness each week. The content for 8 weeks would include knowledge about depression, recognition of depression and depressive mood, symptom management, adaptation skills and coping skills, myths of depression, depression prevention, and referral information for mental health.

The investigators would evaluate the effectiveness of the two groups using the outcome assessment of BDI-II, WHOQOL-BREF, BAI, OSA, and COPM 1 week before intervention (pre-test) and 1 week after intervention (post-test).

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 and 25
* Has Beck Depression Inventory-2 (BDI-II) score of at least mild severity, with no upper limit
* Able to communicate through LINE app
* Able to read Chinese and willing to participate in research

Exclusion Criteria:

* Meets the Diagnostic and Statistical Manual of Mental Disorders-V, such as schizophrenia, substance abuse, and Bipolar disorder
* Has ever been diagnosed as any significant physical illness, such as cancer, organ damage, and stroke
* Refuse to be assigned to different groups randomly

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Ling Chen, Doctor, Study Director — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ritvo P, Knyahnytska Y, Pirbaglou M, Wang W, Tomlinson G, Zhao H, Linklater R, Bai S, Kirk M, Katz J, Harber L, Daskalakis Z. Online Mindfulness-Based Cognitive Behavioral Therapy Intervention for Youth With Major Depressive Disorders: Randomized Controlled Trial. J Med Internet Res. 2021 Mar 10;23(3):e24380. doi: 10.2196/24380. PMID 33688840
- [Result] Hofmann SG, Smits JA. Cognitive-behavioral therapy for adult anxiety disorders: a meta-analysis of randomized placebo-controlled trials. J Clin Psychiatry. 2008 Apr;69(4):621-32. doi: 10.4088/jcp.v69n0415. PMID 18363421
- [Result] Baker F, Intagliata J. Quality of life in the evaluation of community support systems. Eval Program Plann. 1982;5(1):69-79. doi: 10.1016/0149-7189(82)90059-3. PMID 10257372
- [Result] Simmons S. Quality of life in community mental health care--a review. Int J Nurs Stud. 1994 Apr;31(2):183-93. doi: 10.1016/0020-7489(94)90044-2. PMID 8206699
- [Result] Solis AC, Lotufo-Neto F. Predictors of quality of life in Brazilian medical students: a systematic review and meta-analysis. Braz J Psychiatry. 2019 Nov-Dec;41(6):556-567. doi: 10.1590/1516-4446-2018-0116. PMID 30994854
- [Result] Gan GG, Yuen Ling H. Anxiety, depression and quality of life of medical students in Malaysia. Med J Malaysia. 2019 Feb;74(1):57-61. PMID 30846664
- [Result] Surawy C, McManus F, Muse K, Williams JM. Mindfulness-Based Cognitive Therapy (MBCT) for Health Anxiety (Hypochondriasis): Rationale, Implementation and Case Illustration. Mindfulness (N Y). 2015;6(2):382-392. doi: 10.1007/s12671-013-0271-1. PMID 25798209
- [Result] Fjorback LO, Arendt M, Ornbol E, Fink P, Walach H. Mindfulness-based stress reduction and mindfulness-based cognitive therapy: a systematic review of randomized controlled trials. Acta Psychiatr Scand. 2011 Aug;124(2):102-19. doi: 10.1111/j.1600-0447.2011.01704.x. Epub 2011 Apr 28. PMID 21534932
- [Result] Joyce S, Shand F, Tighe J, Laurent SJ, Bryant RA, Harvey SB. Road to resilience: a systematic review and meta-analysis of resilience training programmes and interventions. BMJ Open. 2018 Jun 14;8(6):e017858. doi: 10.1136/bmjopen-2017-017858. PMID 29903782
- [Result] Luo Y, Xia W, Cheung AT, Ho LLK, Zhang J, Xie J, Xiao P, Li HCW. Effectiveness of a Mobile Device-Based Resilience Training Program in Reducing Depressive Symptoms and Enhancing Resilience and Quality of Life in Parents of Children With Cancer: Randomized Controlled Trial. J Med Internet Res. 2021 Nov 29;23(11):e27639. doi: 10.2196/27639. PMID 34847060
- [Result] Guardino CM, Dunkel Schetter C, Bower JE, Lu MC, Smalley SL. Randomised controlled pilot trial of mindfulness training for stress reduction during pregnancy. Psychol Health. 2014;29(3):334-49. doi: 10.1080/08870446.2013.852670. Epub 2013 Nov 1. PMID 24180264
- [Result] Lau N, O'Daffer A, Colt S, Yi-Frazier JP, Palermo TM, McCauley E, Rosenberg AR. Android and iPhone Mobile Apps for Psychosocial Wellness and Stress Management: Systematic Search in App Stores and Literature Review. JMIR Mhealth Uhealth. 2020 May 22;8(5):e17798. doi: 10.2196/17798. PMID 32357125
- [Result] Uthman OA, Nduka CU, Abba M, Enriquez R, Nordenstedt H, Nalugoda F, Kengne AP, Ekstrom AM. Comparison of mHealth and Face-to-Face Interventions for Smoking Cessation Among People Living With HIV: Meta-Analysis. JMIR Mhealth Uhealth. 2019 Jan 7;7(1):e203. doi: 10.2196/mhealth.9329. PMID 30617044
- [Result] Josephine K, Josefine L, Philipp D, David E, Harald B. Internet- and mobile-based depression interventions for people with diagnosed depression: A systematic review and meta-analysis. J Affect Disord. 2017 Dec 1;223:28-40. doi: 10.1016/j.jad.2017.07.021. Epub 2017 Jul 10. PMID 28715726
- [Result] Zhang MW, Ho RC. Moodle: The cost effective solution for internet cognitive behavioral therapy (I-CBT) interventions. Technol Health Care. 2017;25(1):163-165. doi: 10.3233/THC-161261. No abstract available. PMID 27689560
- [Result] Sun Y, Li Y, Wang J, Chen Q, Bazzano AN, Cao F. Effectiveness of Smartphone-Based Mindfulness Training on Maternal Perinatal Depression: Randomized Controlled Trial. J Med Internet Res. 2021 Jan 27;23(1):e23410. doi: 10.2196/23410. PMID 33502326
- [Result] Pan AW, Chung L, Hsin-Hwei G. Reliability and validity of the Canadian Occupational Performance Measure for clients with psychiatric disorders in Taiwan. Occup Ther Int. 2003;10(4):269-77. doi: 10.1002/oti.190. PMID 14647540
- [Result] Winnebeck E, Fissler M, Gartner M, Chadwick P, Barnhofer T. Brief training in mindfulness meditation reduces symptoms in patients with a chronic or recurrent lifetime history of depression: A randomized controlled study. Behav Res Ther. 2017 Dec;99:124-130. doi: 10.1016/j.brat.2017.10.005. Epub 2017 Oct 12. PMID 29078199
- See also: World Health Organization(2021).Depression. — https://www.who.int/news-room/fact-sheets/detail/depression
- See also: 社團法人臺灣憂鬱症防治協會（2021）。青少年憂鬱防治與心理健康促進：需要你我共同參與。 — https://www.depression.org.tw/knowledge/info.asp?/97.html
- See also: 台灣人類職能模式研究與應用發展中心-職能治療(MOHO center in Taiwan)(2009)。職能自我評估-中文版。 — http://mohocentertaiwan.blogspot.com/2009/02/blog-post_9504.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: dates of the recruitment period：2022/02/14~2022/03/14 recruitment location: School website or Online platform
Pre-assignment Details: Participants who (1) have a psychiatric diagnosis, (2) are currently receiving counseling, (3)are not from the medical university in Taiwan, and (4) are unwilling to participate in the study will be excluded.
Groups:
- online mindfulness-based cognitive therapy program: The online mindfulness-based cognitive program was delivered on the platform of LINE to the experimental group 3 times a week for 8 weeks mindfulness-based cognitive therapy, which were detailed mindfulness-based skills training with pictures or short videos, techniques application in different scenarios, and concepts consolidation through a web-based assignment.
Period: Overall Study
Arm/Group | online mindfulness-based cognitive therapy program | mental health education
Started | 26 | 26
Completed | 23 | 23
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Online Mindfulness-based Cognitive Therapy Program: The online mindfulness-based cognitive program was delivered on the platform of LINE to the experimental group 3 times a week for 8 weeks, which were detailed mindfulness-based skills training with pictures or short videos, techniques application in different scenarios, and concepts consolidation through a web-based assignment.
- Total: Total of all reporting groups
Arm/Group | Online Mindfulness-based Cognitive Therapy Program | Mental Health Education | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.88 (1.56) | 21.92 (1.02) | 21.40 (0.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 39
  Male | 9 | 4 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Departments [Count of Participants; unit: Participants]
  Department of Occupational Therapy | 11 | 7 | 18
  Department of Speech Language Pathology and Audiology | 5 | 7 | 12
  Department of Nursing | 2 | 1 | 3
  Department of Nutrition | 1 | 3 | 4
  Department of Public Health | 1 | 2 | 3
  School of Medicine | 0 | 2 | 2
  Department of Physical Therapy | 1 | 1 | 2
  Department of Medical Sociology and Social Work | 0 | 1 | 1
  Department of Medical Laboratory and Biotechnology | 1 | 0 | 1
  Department of Medical Imaging and Radiological Sciences | 1 | 0 | 1
  Department of Health Industry Technology Management | 1 | 1 | 2
  Department of Medical Informatics | 1 | 1 | 2
  Department of Applied Foreign Languages | 1 | 0 | 1
Grades [Count of Participants; unit: Participants]
  freshman | 3 | 0 | 3
  sophomore | 5 | 4 | 9
  junior | 9 | 8 | 17
  senior | 9 | 12 | 21
  sixth year of undergraduate school | 0 | 2 | 2
Course units [Mean (Standard Deviation); unit: units] | 17.12 (5.59) | 15.34 (4.94) | 16.23 (0.74)
Clubs [Count of Participants; unit: Participants]
  Yes | 6 | 6 | 12
  No | 20 | 20 | 40
Part-time jobs [Count of Participants; unit: Participants]
  Yes | 10 | 10 | 20
  No | 16 | 16 | 32
Livings status [Count of Participants; unit: Participants]
  Living with classmates/friends | 9 | 11 | 20
  Living alone | 10 | 6 | 16
  Living with family/relatives | 5 | 8 | 13
  other | 2 | 1 | 3
Economic status [Count of Participants; unit: Participants]
  Family allowance | 23 | 23 | 46
  Self-sufficient | 1 | 1 | 2
  Family allowance + Self-sufficiency | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: BDI-II -Pretest
Description: The Beck Depression Inventory II (BDI-II) is a 21-item self-report questionnaire designed to measure the level of severity of disorders of depression. Items are scored from 0 to 3; higher scores indicate greater symptom severity. In the BDI-II values below 13 points are regarded as no or minimal depressive symptoms. Values between 14 and 19 points indicate a mild expression of depressive symptoms, values between 20 and 28 points a moderate severity. Scores between 29 and 63 are regarded as evidence of severe depressive disorder.
Time Frame: BDI-II score at pre-test (1week before intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | online mindfulness-based cognitive therapy program | mental health education
Number analyzed (Participants) | 23 | 23
score on a scale | 12.54 (10.31) | 14.42 (11.5)

2. Primary Outcome: BDI-II -Posttest
Description: as for outcome 1
Time Frame: 1 week after the intervention, corresponding to Week 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | online mindfulness-based cognitive therapy program | mental health education
Number analyzed (Participants) | 23 | 23
score on a scale | 7 (7.83) | 9.87 (10.1)

3. Primary Outcome: WHOQOL-BREF-TW -Pretest
Description: The World Health Organization Quality-of-Life Scale (WHOQOL-BREF) is a 28-item self-report questionnaire with a five point rating scale for each item (from 1 to 5). There are four domains in WHOQOL-BREF, including physical health, psychological health, social relationships, and environment. The Physical Health domain consists of 7 items, with a total score range of 7 to 35; the Psychological domain includes 6 items, ranging from 6 to 30; the Social Relationships domain comprises 4 items, with scores ranging from 4 to 20; and the Environment domain contains 9 items, with a range of 9 to 45.
  Two additional items are assessed separately: Question 1 evaluates an individual's overall perception of quality of life, while Question 2 assesses their overall perception of health. Each of these two items is scored on a scale from 1 to 5.
  Domain scores are scaled in a positive direction, meaning that higher scores indicate better quality of life in the corresponding domain.
Time Frame: WHOQOL-BREF-TW score at pre-test (1week before intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | online mindfulness-based cognitive therapy program | mental health education
Number analyzed (Participants) | 23 | 23
score on a scale
  Overall quality of Life | 3.38 (0.75) | 3.15 (0.73)
  General Health facet | 2.88 (0.59) | 2.65 (0.75)
  Physical Health | 26.31 (3.96) | 23.85 (4.4)
  Psychological | 18.38 (4.73) | 17.81 (4.11)
  Social relationships | 14.54 (2.79) | 13.96 (1.95)
  Environment | 33.81 (4.54) | 32 (4.72)

4. Primary Outcome: WHOQOL-BREF-TW -Posttest
Description: as for outcome 3
Time Frame: 1 week after the intervention, corresponding to Week 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | online mindfulness-based cognitive therapy program | mental health education
Number analyzed (Participants) | 23 | 23
score on a scale
  Overall quality of Life | 3.87 (0.69) | 3.48 (0.73)
  General Health facet | 3.04 (1.02) | 3.13 (0.92)
  Physical Health | 28.13 (4.32) | 25.74 (3.6)
  Psychological | 21.13 (5.15) | 18.7 (3.76)
  Social relationships | 15.52 (2.5) | 14.7 (2.18)
  Environment | 36.39 (5.32) | 32.61 (4.52)

5. Secondary Outcome: BAI -Pretest
Description: The Beck Anxiety Inventory (BAI) is a 21-item self-report measure designed to reflect the severity of somatic and cognitive symptoms of anxiety over the previous week. Items are scored from 0 to 3; higher scores indicate greater symptom severity. The BAI scores are classified as minimal anxiety (0 to 7), mild anxiety (8 to 15), moderate anxiety (16 to 25), and severe anxiety (30 to 63).
Time Frame: BAI score at pre-test (1week before intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | online mindfulness-based cognitive therapy program | mental health education
Number analyzed (Participants) | 26 | 26
score on a scale | 9.31 (7.36) | 8.65 (7.65)

6. Secondary Outcome: BAI -Posttest
Description: as for outcome 5
Time Frame: 1 week after the intervention, corresponding to Week 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | online mindfulness-based cognitive therapy program | mental health education
Number analyzed (Participants) | 23 | 23
score on a scale | 5.52 (7.38) | 6.52 (6.71)

7. Secondary Outcome: OSA -Pretest
Description: The Occupational Self-Assessment (OSA) evaluates self-perceived occupational competence and environmental support. The questionnaire includes two sections: Self-Competence and Environment. The Self-Competence section has 21 items divided into three subscales-Skills/Performance (11 items), Habituation (5 items), and Volition (5 items)-and the Environment section has 8 items assessing perceived environmental support. Each item is rated on a 4-point scale, where 1 indicates the lowest and 4 the highest level of perceived competence or support. The possible score ranges are 11-44 for Skills/Performance, 5-20 for Habituation, 5-20 for Volition, and 8-32 for Environment. Higher scores represent greater self-perceived occupational competence and stronger environmental support.
Time Frame: OSA score at pre-test (1week before intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | online mindfulness-based cognitive therapy program | mental health education
Number analyzed (Participants) | 26 | 26
score on a scale
  Skills/Performance | 33.62 (4.73) | 30.73 (4.62)
  Habituation | 14.42 (2.76) | 12.96 (2.81)
  Volition | 13.88 (2.63) | 12.69 (2.9)
  Environment | 27.42 (3.7) | 26.65 (3.82)

8. Secondary Outcome: OSA -Posttest
Description: as for outcome 7
Time Frame: 1 week after the intervention, corresponding to Week 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | online mindfulness-based cognitive therapy program | mental health education
Number analyzed (Participants) | 23 | 23
score on a scale
  Skills/Performance | 35.3 (4.99) | 32.65 (4.46)
  Habituation | 16.35 (2.74) | 13.83 (2.37)
  Volition | 15.96 (2.85) | 14.04 (3.31)
  Environment | 28.7 (3.78) | 26.96 (4.37)

9. Secondary Outcome: COPM -Pretest
Description: The Canadian Occupational Performance Measure (COPM) is an individualized measure designed for use by occupational therapists to detect self-perceived change in occupational performance problems over time. The therapist calculates an average COPM performance score and satisfaction score. These typically range between 1 and 10, where 1 indicates poor performance and low satisfaction, respectively, while 10 indicates very good performance and high satisfaction.
Time Frame: COPM score at pre-test (1week before intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | online mindfulness-based cognitive therapy program | mental health education
Number analyzed (Participants) | 26 | 26
score on a scale
  Performance | 5.93 (1.51) | 4.62 (1.46)
  Satisfaction | 5.39 (1.84) | 4.22 (1.77)

10. Secondary Outcome: COPM -Posttest
Description: as for outcome 9
Time Frame: 1 week after the intervention, corresponding to Week 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | online mindfulness-based cognitive therapy program | mental health education
Number analyzed (Participants) | 23 | 23
score on a scale
  Performance | 7.03 (1.65) | 6.01 (1.37)
  Satisfaction | 6.85 (1.85) | 6.06 (1.66)

ADVERSE EVENTS:
Time Frame: From intervention initiation to post-intervention follow-up for each participant, up to 19 weeks.
Description: This research involved participatory mindfulness practice and questionnaire surveys, without using invasive measures. Throughout the entire study period, from intervention initiation to post-intervention follow-up (April 20, 2023 to September 1, 2023), no risks, harms, or adverse events occurred to participants.
Groups:
- online mindfulness-based cognitive therapy program: The online mindfulness-based cognitive program was delivered on the platform of LINE to the experimental group 3 times a week for 8 weeks mindfulness-based cognitive therapy: Participants in the experimental group would be arranged to attend online mindfulness-based cognitive programs for eight weeks. Each week was divided into 3 parts, which were detailed mindfulness-based skills training with pictures or short videos, techniques application in different scenarios, and concepts consolidation through a web-based assignment.
Arm/Group | online mindfulness-based cognitive therapy program | mental health education
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT05804877/Prot_SAP_ICF_000.pdf